CLINICAL TRIAL: NCT03451617
Title: Randomized Clinical Evaluation of Alpine® vs. Xpedition® Stent Delivery System of the XIENCE® Everolimus-eluting Stent
Brief Title: Alpine vs. Xpedition: Evaluation of Stent Delivery System
Acronym: AXES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Groningen (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Pim van der Harst, Prof. Dr. P. van der Harst, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201600966
Record Dates: First submitted 2017-11-09; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xpedition stent delivery system (Other)
  Interventions: Device: Stent delivery with Xpedition
- Alpine stent delivery system (Other)
  Interventions: Device: Stent delivery with Alpine

INTERVENTIONS:
Device: Stent delivery with Xpedition — Use of Xpedition stent delivery system to implant the XIENCE stent
  Arms: Xpedition stent delivery system
Device: Stent delivery with Alpine — Use of Alpine stent delivery system to implant the XIENCE stent
  Arms: Alpine stent delivery system

SUMMARY:
To evaluate and compare the performance of two stent delivery systems for percutaneous coronary intervention with everolimus-eluting stent.

DETAILED DESCRIPTION:
Rationale: The current gold standard for percutaneous coronary intervention (PCI) is the second generation drug-eluting stent (DES). The most commonly used DES is the everolimus-eluting stent (EES). New stent delivery systems for PCI with EES are developed to optimize strength, flexibility and pushability of the catheter. The effect on procedural time of new stent delivery systems has not yet been investigated in clinical practice.

Objective: To evaluate and compare the performance of two stent delivery systems for PCI with EES.

Study design: Randomized comparative trial with 500 patients in the University Medical Center Groningen (UMCG).

Study population: All patients undergoing PCI with EES, aged 18 years or older, will be considered for eligibility. Patients will be excluded when scheduled for chronic total occlusion (CTO) PCI or if verbal informed consent cannot be obtained.

Intervention: The first group will undergo PCI with the XIENCE EES using the Alpine stent delivery system, the second group will undergo PCI with the Xpedition stent delivery system.

Main study parameters/endpoints: The primary endpoint is the proportion of procedures with crossing time (from introduction of guidewire to stent deployment) longer than 30 minutes. Secondary endpoints include procedural time (from heparin administration to removal of catheter sheath, mins), use of additional materials, total procedural costs, radiation dose (μGym2), radiation time (mins), and contrast dose (ml).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing PCI with EES, aged 18 years or older

Exclusion Criteria:

* Chronic total occlusion (CTO) PCI
* Inability to obtain (verbal) informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-10-05 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Crossing time | During PCI procedure
  Proportion of procedures with crossing time (from introduction of guidewire to stent deployment) longer than 30 minutes.

SECONDARY OUTCOMES:
Procedural time | During PCI procedure
Total procedural costs | During PCI procedure
  Total cost of the materials used during the procedure (stent delivery system and additional materials) in euros.
Radiation dose | During PCI procedure
Radiation time | During PCI procedure
Contrast dose | During PCI procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided